CLINICAL TRIAL: NCT05054634
Title: Psycho-oncological Intervention Through Counselling in Patients With Differentiated Thyroid Cancer in Treatment With Radioiodine: A Non-randomized Controlled Study
Brief Title: Psycho-oncological Intervention Through Counselling in Patients With Differentiated Thyroid Cancer in Treatment With Radioiodine
Acronym: COUNTHY
Status: Completed | Type: Observational
Sponsor: Quironsalud (Other)
Responsible Party: Principal Investigator, Manuel Sureda Gonzalez, Principal Investigator, Quironsalud
Other Study IDs: COUNTHY
Record Dates: First submitted 2021-09-03; First posted 2021-09-23 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Thyroid Cancer
Keywords: cancer; oncology; psycho-oncology; psychotherapy; thyroid cancer; radioisotope therapy; quality of life
MeSH Terms: conditions — Thyroid Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental Group (EG): Patients diagnosed with DTC, treated with thyroidectomy and candidates to RIT to be treated in Nuclear Medicine (NM) Service of Hospital Quirónsalud Torrevieja were considered to be included in the study. They were alternatively assigned to the EG or CG, according to their order of entry.
  Interventions: Behavioral: Psycho-oncological Intervention Based on Counselling (PIBC)
- Control Group (CG): Patients diagnosed with DTC, treated with thyroidectomy and candidates to RIT to be treated in Nuclear Medicine (NM) Service of Hospital Quirónsalud Torrevieja were considered to be included in the study. They were alternatively assigned to the EG or CG, according to their order of entry.

INTERVENTIONS:
Behavioral: Psycho-oncological Intervention Based on Counselling (PIBC) — Patients in EG received a psycho-oncological intervention based on Counselling (PIBC) following the scheme proposed by Arranz and Cancio in addition to the standard treatment. The evolution of anxiety and depression was evaluated using Hospital Anxiety and Depression Scale (HADS). The aim of the study was to evaluate the effectiveness of a PIBC in reducing anxiety and depression of patients with DTC. Other QoL relevant items were also evaluated using the Short Form-36 Health Survey (SF-36) and Psychological General Well-Being Index (PGWBI) scales.
  Groups: Experimental Group (EG)

SUMMARY:
Diagnosis and treatment of differentiated thyroid carcinomas cause anxiety and depression. Additionally, these patients suffer hormonal alterations, associated with psychological symptoms (changes in mood, emotional instability, memory loss, etc.). This study aims to evaluate the effectiveness of a psycho-oncological intervention based on Counselling to reduce anxiety and depression related with the treatment in patients with differentiated thyroid carcinomas.

DETAILED DESCRIPTION:
A non-randomized controlled study, with two groups (experimental, n=37, and control, n=38) and baseline and post-treatment measures was designed. Patients in experimental group received a psycho-oncological intervention based on Counselling in addition to the standard treatment. The independent variable was the assigned group and the dependent one was the evolution of anxiety and depression, analyzed separately, both evaluated using HADS. Other relevant covariables related with quality of life were also analyzed using SF-36 and PGWBI scales.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with DTC (differentiated thyroid carcinoma)
* Initial treatment by total thyroidectomy
* Treatment with RIT after physiological stimulation of thyroid-stimulating hormone (TSH) by suppression of hormone replacement therapy (HRT) for a month
* Fluid Spanish speaker
* 18 years or over
* Obtaining informed consent

Exclusion Criteria:

* Diagnosis or treatment for psychiatric disorders
* Any type of illness with serious impact in medical condition
* Inability to communicate or to process the information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Between June 2013 and September 2014, a total of 75 patients were included in the study, 37 in the EG (Experimental Group) and 38 in the CG (Control Group). No patient declined to be included. No statistically significant differences were observed in sociodemographic characteristics between both groups.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2013-06-01 (Actual); Primary Completion 2014-09-30 (Actual); Study Completion 2015-03-31 (Actual)

PRIMARY OUTCOMES:
Anxiety and depression of patients with DTC (Differentiated Thyroid Carcinoma) after a PIBC (Psycho-oncological intervention based on Counselling). | Through study completion, an average of 2 months
  Research on the effectiveness of psycho-oncological interventions in the last 20 years has been classified according to the phase of the oncological process and to the objectives to be achieved. According to the objectives, the interventions focuses on controlling the symptoms associated with the disease, on improving the emotional state, on improving and recover the functional status of patients and on improving quality of life (QoL).
  Anxiety and depression were evaluated through the HADS scale [Zigmond et al. 1983, Herrmann 1997]. A minimum goal of 3-point reduction in the HADS scale was considered as an improvement. Effect size measure was calculated with Cohen's d for the difference between EG and CG in the primary outcome variable at post-treatment, for both anxiety and depression.
Quality of Life of patients with DTC (Differentiated Thyroid Carcinoma) after a PIBC (Psycho-oncological intervention based on Counselling). | Through study completion, an average of 2 months
  The Quality of Life was measured through the SF-36 questionnaire [Vilagut G et al 2005, Molina RT 2005, Martin M 2004].
Mood, perceived well-being and emotional impact of patients with DTC (Differentiated Thyroid Carcinoma) after a PIBC (Psycho-oncological intervention based on Counselling). | Through study completion, an average of 2 months
  Those variables were measured through the PGWBI of Dupuy [Vilagut G et al 2005, Molina RT 2005, Martin M 2004].

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Sureda, MD, Study Chair — Plataforma de Oncología. Hospital Quironsalud Torrevieja
Locations (1):
- Hospital Quironsalud Torrevieja, Torrevieja, Spain